CLINICAL TRIAL: NCT02119650
Title: A Randomized, Double-Blind Phase 2 Study of Ruxolitinib or Placebo in Combination With Pemetrexed/Cisplatin and Pemetrexed Maintenance for Initial Treatment of Subjects With Nonsquamous Non-Small Cell Lung Cancer That Is Stage IIIB, Stage IV, or Recurrent
Brief Title: Ruxolitinib in Combination With Pemetrexed/Cisplatin in Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated as other related studies of ruxolitinib did not provide sufficient efficacy to warrant continuation.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-266
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: NSCLC (Non-small Cell Lung Carcinoma)
Keywords: Non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ruxolitinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruxolitinib plus Pemetrexed/Cisplatin (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Pemetrexed; Drug: Cisplatin
- Placebo plus Pemetrexed/Cisplatin (Active Comparator)
  Interventions: Drug: Placebo; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets to be administered by mouth at dose selected from safety run-in phase (Ruxolitinib 15 mg twice daily (BID))
  Other Names: Jakafi ®; Jakavi ®
  Arms: Ruxolitinib plus Pemetrexed/Cisplatin
Drug: Placebo — 5 mg matching placebo tablets to be administered by mouth
  Arms: Placebo plus Pemetrexed/Cisplatin
Drug: Pemetrexed — 500 mg/m^2 administered as an intravenous infusion over 10 minutes
  Other Names: Alimta®
Drug: Cisplatin — 75 mg/m^2 infused over 2 hours beginning 30 ± 5 minutes after the end of the pemetrexed infusion

SUMMARY:
The purpose of this study was to determine if ruxolitinib, in combination with Pemetrexed/Cisplatin and Pemetrexed Maintenance, is safe and effective in the treatment of nonsquamous non-small cell lung cancer (NSCLC) that is Stage IIIB, Stage IV, or recurrent.

DETAILED DESCRIPTION:
The study consisted of an open-label, safety run-in (consisting of 1 to 4 cohorts of 9 participants each), to confirm the safety of ruxolitinib in combination with pemetrexed/cisplatin in participants with nonsquamous non-small cell lung cancer (NSCLC) that is Stage IIIB, Stage IV, or recurrent. Participants in the safety run-in received open-label ruxolitinib and pemetrexed and cisplatin.

In the second part of the study, participants enrolled and randomized and received pemetrexed and cisplatin (open-label) and either ruxolitinib or placebo in a blinded manner. The dose of ruxolitinib administered was determined from the data produced in the safety run-in phase.

Treatment consisted of repeating 21-day cycles. Participants received infusions of pemetrexed and cisplatin on Day 1 of each cycle and ruxolitinib/placebo was self-administered during the entire cycle. Maintenance therapy with ruxolitinib or placebo in combination with pemetrexed, based on the original treatment assignment, was allowed for participants eligible for maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of nonsquamous NSCLC that is Stage IIIB Stage IV, or recurrent after prior definitive intervention (radiation, surgery, or chemoradiation therapy, with or without adjuvant or neoadjuvant chemotherapy).
* Radiographically measurable or evaluable disease.
* Life expectancy of at least 12 weeks.
* Tumor without activating driver mutations for which there is available therapy (eg, tumor without mutations in epidermal growth factor receptor or anaplastic lymphoma).
* An modified Glasgow Prognostic Score (mGPS) of 1 or 2 as defined below:

  * Criteria:

    * C-reactive protein >10 mg/L AND albumin ≥35 g/L; Score = 1
    * C-reactive protein >10 mg L AND albumin <35 g/L; Score = 2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Adequate renal, hepatic, and bone marrow function demonstrated by protocol-specified laboratory parameters at the screening visit.

Exclusion Criteria:

* Squamous or mixed histology (eg, adenosquamous) NSCLC
* Previous systemic therapy for advanced or metastatic disease.
* Known active central nervous system (CNS) metastases.
* Current or previous other malignancy within 2 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy without sponsor approval.
* Current uncontrolled cardiac disease such as angina or myocardial infarction, congestive heart failure including New York Heart Association functional classification of 3, or arrhythmia requiring treatment.
* Uncontrolled concomitant medical conditions, including, but not limited to, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2016-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard T Kennealey, MD, Study Director — Incyte Corporation
Locations (30):
- United States (30):
  - Phoenix, Arizona
  - Fayetteville, Arkansas
  - Fresno, California
  - La Jolla, California
  - San Diego, California
  - San Francisco, California
  - Lone Tree, Colorado
  - Norwich, Connecticut
  - Southington, Connecticut
  - Augusta, Georgia
  - Joliet, Illinois
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Kansas City, Kansas
  - Detroit, Michigan
  - St Louis, Missouri
  - Reno, Nevada
  - Lebanon, New Hampshire
  - Mount Kisco, New York
  - New York, New York
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Portland, Oregon
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Ogden, Utah
  - Leesburg, Virginia
  - Kennewick, Washington
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 42 study centers (25 in the United States, 4 in Spain, 3 in France, 3 in Portugal, 2 in Denmark, 2 in Germany, 2 in Italy, 1 in the Netherlands).
Groups:
- Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin: Ruxolitinib was self-administered as a 15 mg twice daily (BID) oral treatment during the randomized, double-blind treatment, without regard to food. Pemetrexed 500 mg/m^2 was administered as an intravenous infusion over 10 minutes, and 75 mg/m^2 Cisplatin was infused over 2 hours beginning 30 ± 5 minutes after the end of the pemetrexed infusion on Day 1 of each 21-day cycle (Treatment Cycles).
- Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin: Matching placebo was self-administered as a 15 mg BID oral treatment during the randomized, double-blind treatment, without regard to food. Pemetrexed 500 mg/m^2 was administered as an intravenous infusion over 10 minutes, and 75 mg/m^2 Cisplatin was infused over 2 hours beginning 30 ± 5 minutes after the end of the pemetrexed infusion on Day 1 of each 21-day cycle (Treatment Cycles).
Period: Overall Study
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Started | 39 | 37
Completed | 14 (Participants with treatment ongoing when the study was terminated.) | 11 (Participants with treatment ongoing when the study was terminated.)
Not Completed | 25 | 26
Not completed — Adverse Event | 3 | 4
Not completed — Subject decision | 2 | 3
Not completed — Disease progression | 11 | 14
Not completed — Death | 5 | 1
Not completed — Noncompliance with study treatment | 1 | 1
Not completed — Study terminated by the sponsor | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Multiple reasons for termination | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of participants that were randomized in the study.
Groups:
- Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin: Ruxolitinib was self-administered as a 15 mg BID oral treatment during the randomized, double-blind treatment, without regard to food. Pemetrexed 500 mg/m^2 was administered as an intravenous infusion over 10 minutes, and 75 mg/m^2 Cisplatin was infused over 2 hours beginning 30 ± 5 minutes after the end of the pemetrexed infusion on Day 1 of each 21-day cycle (Treatment Cycles).
- Total: Total of all reporting groups
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.85) | 62.0 (8.55) | 61.8 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 24 | 23 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 36 | 33 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.67 (6.402) | 27.65 (7.26) | 27.66 (6.787)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death due to any cause. Participants without death observed at the time of the analysis were censored at last date known to be alive. The median overall survival time was estimated using the Kaplan-Meier method. Overall survival was compared between treatment groups using log-rank test.
Time Frame: Randomization until death due to any cause; up to 16 months or data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of participants that were randomized in the study.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 37
months | 7.5 [5.7 to NA] — Not evaluable due to insufficient number of participants with events. | 5.9 [4.0 to NA] — Not evaluable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin vs Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin; Test type: Other; p = 0.7562, Log Rank; The 2-sided p-value was calculated based on the log-rank test and stratified by modified Glasgow Prognostic Score (mGPS); Hazard Ratio (HR) = 0.877, 80% CI 2-sided [0.509 to 1.51]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization until the earliest date of disease progression determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause if sooner. Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum Longest Diameter (LD) recorded since the treatment started or the appearance of one or more new lesions, unequivocal progression of non-target lesions or increase in disease burden for subjects with only nonmeasurable disease.
Time Frame: Randomization to disease progression, or death due to any cause if sooner; up to 16 months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of participants that were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 37
Months | NA [NA to NA] — Progression-free Survival (PFS) was not conducted due to early termination of the study and insufficient number of participants with events. | NA [NA to NA] — Progression-free Survival (PFS) was not conducted due to early termination of the study and insufficient number of participants with events.

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate determined by radiographic disease assessments per RECIST (v1.1), by investigator assessment and was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST) at any post baseline visit. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) : Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Baseline through end of study; up to 16 months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of participants that were randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 37
Participants
  Overall Response | 12 | 13
  Complete Response | 0 | 0
  Partial Response | 12 | 13
  Stable Disease | 4 | 5
  Progressive Disease | 6 | 4
  Unable to Evaluate | 2 | 3
  Not Assessed | 15 | 12

4. Secondary Outcome: Duration of Response
Description: For objective responders, the duration of response is defined as the difference of the end of response and the start of response. The start of a response was the first visit where the subject achieves PR or better based on RECIST v1.1 criteria. The end of response was the first visit after PD based on RECIST v1.1 criteria.
Time Frame: From the start of response to the end of response; up to 16 months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of participants that were randomized in the study.
Measure: Median (80% Confidence Interval); unit: weeks
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Number analyzed (Participants) | 12 | 13
weeks | 20.14 [18.00 to 30.71] | 12.14 [6.00 to 24.00]

5. Secondary Outcome: Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A treatment-emergent AE was defined as an event occurring (or worsening of any pre-existing) after exposure to at least 1 dose of study drug. A treatment-related AE was defined as an event with a definite, probable, or possible causality to study medication. A serious AE is an event resulting in death, hospitalization, persistent or significant disability/incapacity, or is life threatening, a congenital anomaly/birth defect or requires medical or surgical intervention to prevent 1 of the outcomes above. The intensity of an AE was graded according to the National Cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 4.03: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (life-threatening).
Time Frame: Baseline through approximately 30 days post treatment discontinuation; up to 16 months or to the data cutoff 11FEB2016.
Population: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 37
Participants
  Participants who had any TEAEs | 39 | 36
  Participants who had treatment-related TEAEs | 16 | 28
  Participants with any serious TEAE | 19 | 16
  Participants who had Grade 3 or higher TEAEs | 25 | 22
  Participants with a fatal TEAE | 4 | 4
  TEAEs related to reference therapy | 30 | 35
  Participants who were hospitalized due to TEAEs | 16 | 15
  Participants who discontinued drug due to TEAEs | 2 | 4
  Participants who interrupted drug due to TEAEs | 11 | 15
  Discontinued reference therapy due to TEAEs | 4 | 7
  Interrupted reference therapy due to TEAEs | 8 | 7
  Participants given concomitant meds due to TEAEs | 36 | 32
  Procedure/nondrug therapy due to TEAEs | 17 | 12

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through approximately 30 days post treatment discontinuation; up to 16 months or to the data cutoff 11FEB2016.
Description: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug.
Arm/Group | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin
Serious Adverse Events (participants affected / at risk) | 19/39 | 16/37
Other Adverse Events (participants affected / at risk) | 37/39 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin (N=39) | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin (N=37)
Pneumonia (Infections and infestations) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
VIth nerve disorder (Nervous system disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment: Ruxolitinib + Pemetrexed/Cisplatin (N=39) | Double-Blind Treatment: Placebo Plus Pemetrexed/Cisplatin (N=37)
Anaemia (Blood and lymphatic system disorders) | 15 | 12
Neutropenia (Blood and lymphatic system disorders) | 8 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 13 | 13
Diarrhoea (Gastrointestinal disorders) | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Dysphagia (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 20 | 32
Stomatitis (Gastrointestinal disorders) | 10 | 7
Vomiting (Gastrointestinal disorders) | 7 | 12
Chest pain (General disorders) | 3 | 2
Fatigue (General disorders) | 13 | 14
Oedema peripheral (General disorders) | 8 | 5
Pyrexia (General disorders) | 7 | 4
Candida infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
Blood calcium decreased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 4 | 2
Weight decreased (Investigations) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 14
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 2 | 6
Dysgeusia (Nervous system disorders) | 2 | 6
Headache (Nervous system disorders) | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Renal failure acute (Renal and urinary disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Hypertension (Vascular disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Ototoxicity (Ear and labyrinth disorders) | 1 | 4
C-reactive protein increased (Investigations) | 1 | 3
Platelet count decreased (Investigations) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthenia (General disorders) | 7 | 12
Malaise (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 3

LIMITATIONS AND CAVEATS:
The study was terminated as other related studies of ruxolitinib did not provide sufficient efficacy to warrant continuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.